CLINICAL TRIAL: NCT03946163
Title: Iraqi Traditional Medicine for Urinary Tract Symptoms: The Effect of Cinnamon on Patients With Chronic Prostatitis/Chronic Pelvic Pain Syndrome; a Pilot Study
Brief Title: The Effect of Cinnamon on Patients With Chronic Prostatitis/Chronic Pelvic Pain Syndrome; a Pilot Study
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Al-Kindy College of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 5 Al-KindyCM
Record Dates: First submitted 2019-05-09; First posted 2019-05-10 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Chronic Prostatitis; Chronic Pelvic Pain Syndrome
Keywords: chronic prostatitis; chronic pelvic pain syndrome; cinnamon; herbal medicine; Traditional medicine

STUDY DESIGN:
Intervention Model Description: The patients will be randomized into two groups, the first group will receive sixty capsules, each capsule contains 1gm of cinnamon bark powder and will be instructed to use it twice daily for one month, the second group will receive 60 capsules containing placebo and will be instructed to use it twice daily for one month
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: the capsules of similar shape, size, color, and smell will be packed in in 60 capsules pack by the preparing pharmacist and labeled as 1 or 2 on the pack, the team will be informed by the content of each pack only after the conclusion of the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- first group (Experimental): each patient will receive sixty capsules, each capsule contained 1gm of cinnamon bark powder and instructed to use it twice daily for one month
  Interventions: Dietary Supplement: cinnamon capsules
- second group (Placebo Comparator): each patient will receive sixty capsules, each capsule contained placebo and instructed to use it twice daily for one month
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Dietary Supplement: cinnamon capsules — each patient will receive sixty capsules, each capsule contained 1gm of cinnamon bark powder and instructed to use it twice daily for one month
  Arms: first group
Drug: Placebo oral capsule — each patient will receive sixty capsules, each capsule contained placebo and instructed to use it twice daily for one month
  Other Names: Placebo
  Arms: second group

SUMMARY:
Chronic prostatitis / chronic pelvic pain syndrome (CP/CPPS) is one of the common urologic problems, nevertheless; its etiology and pathophysiology are poorly understood, with no solid guidelines for effective treatment. The beneficial health attributes of cinnamon and its derivative and components were reported by several researchers, this study is designed to illuminate the possible benefits of cinnamon on patients with Chronic prostatitis / chronic pelvic pain syndrome (CP/CPPS)

DETAILED DESCRIPTION:
Chronic prostatitis / chronic pelvic pain syndrome (CP/CPPS) defined as the "presence of genitourinary pain in the absence of uropathogenic bacteria detected by standard microbiologic methodology" by the National Institutes of Health (NIH) (1) The presence of symptoms resembling that of CP/CPPS in different population fall in the range between 2.2% and 9.7%, with a mean prevalence of 8.2%. making CP/CPPS one of the common urologic problems, nevertheless; its etiology and pathophysiology are poorly understood, with no solid guidelines for effective treatment (2, 3) Prolonged period of antibiotic therapy is usually used as the first line in treatment of CP/CPPS in the first place regardless of the finding of prostatic fluid microscopic examination and culture, when this failed, the next option in management that have been tried and investigated include medications such as alpha-blockers, anti-inflammatory drugs, muscle relaxants, anticonvulsants, or even hormonal manipulation, also physiotherapy, behavioral therapy, herbal or even surgical interventions all have been tried without conclusive evidence supporting the superiority of single treatment option over the others for all patients, making further studying and analysis desirable to get better understanding of the effectiveness of such options or even the trial of different treatment option in the hope of finding effective treatment. (4) Sandalwood (lignum Santali Albi), jasmine, and cinnamon are aromatic herbs that are traditionally used by for regulating qi, removing blood stasis, and relieving pain. (5) Previous studies found cinnamon had an antibacterial effect. (6) Cinnamon is the bark of trees belonging to the genus Cinnamomum. (7) Cinnamon has well known recognizable scent due to its oil content, which has a high concentration of the compound cinnamaldehyde in addition to several other compounds such as cinnamyl acetate, L-borneol, caryophyllene oxide, eugenol, b-caryophyllene, L-bornyl acetate, E-nerolidol, α-terpineol, α-cubebene, terpinolene, and α-thujene. In addition, cinnamon contains a variety of resinous compounds, including cinnamate, cinnamic acid. (8-10) Cinnamon has been long used in kitchens as spice and appetizer without reported serious adverse events. The beneficial health attributes of cinnamon and its derivative and components were reported by several researchers: these include its antimicrobial, anti-inflammatory, antioxidant action, anti-diabetic, and even anticancer actions .nevertheless; further studied are still required to illuminate the potential health benefits of the spice. (11) The National Institutes of Health Chronic Prostatitis Symptoms Index (NIH-CPSI) was developed as a tool to assess the severity of symptoms of CPPS. (12) A reduction of six or more points in NIH-CPSI score is considered clinically perceivable difference by the patients as confirmed by previous studies. (13)

ELIGIBILITY:
Inclusion Criteria:

1. Have symptoms of chronic prostatitis / chronic pelvic pain syndrome
2. Duration of symptoms more than 6 months

Exclusion Criteria:

1. Positive urine culture or positive prostatic secretions culture
2. Food allergies
3. Previous transurethral intervention,
4. Uncontrolled medical disease (such as diabetes, hypertension or asthma),
5. Use of analgesics for other conditions (like musculoskeletal pain or so)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
positive response | 1 month
  A reduction in the NIH-CPSI score of 6 or more points from the initial score

SECONDARY OUTCOMES:
minor positive response | 1 month
  reduction in one or more the sub-scores of the NIH-CPSI

CONTACTS AND LOCATIONS:
Overall Officials: Tawfik J Al-Marzooq, F.I.C.M.S., Principal Investigator — University of Baghdad- Alkindy collage of medicine; Qays A Al-Timimy, F.I.C.M.S., Principal Investigator — University of Baghdad- Alkindy collage of medicine; Harth M Kamber, F.I.C.M.S., Study Director — University of Baghdad- Alkindy collage of medicine; Malath A Hussein, F.I.C.M.S., Principal Investigator — University of Baghdad- Alkindy collage of medicine; Ahmed A Marzouq, F.I.C.M.S., Principal Investigator — University of Baghdad- Alkindy collage of medicine
Locations (1):
- Harth Kamber, Baghdad, (select), Iraq

REFERENCES:
- [Background] Krieger JN, Nyberg L Jr, Nickel JC. NIH consensus definition and classification of prostatitis. JAMA. 1999 Jul 21;282(3):236-7. doi: 10.1001/jama.282.3.236. No abstract available. PMID 10422990
- [Background] Krieger JN, Lee SW, Jeon J, Cheah PY, Liong ML, Riley DE. Epidemiology of prostatitis. Int J Antimicrob Agents. 2008 Feb;31 Suppl 1(Suppl 1):S85-90. doi: 10.1016/j.ijantimicag.2007.08.028. Epub 2007 Dec 31. PMID 18164907
- [Background] Nickel JC. Prostatitis: myths and realities. Urology. 1998 Mar;51(3):362-6. doi: 10.1016/s0090-4295(97)00643-2. PMID 9510337
- [Background] Lee SW. Recent trend of chronic prostatitis/chronic pelvic pain syndrome (CP/CPPS) management. Hanyang Medical Reviews. 2017;37(1):40-6.
- [Background] Hempen C-H, Fischer T. A materia medica for Chinese medicine: plants, minerals, and animal products: Elsevier Health Sciences; 2009.
- [Background] Nabavi SF, Di Lorenzo A, Izadi M, Sobarzo-Sanchez E, Daglia M, Nabavi SM. Antibacterial Effects of Cinnamon: From Farm to Food, Cosmetic and Pharmaceutical Industries. Nutrients. 2015 Sep 11;7(9):7729-48. doi: 10.3390/nu7095359. PMID 26378575
- [Background] Chen P, Sun J, Ford P. Differentiation of the four major species of cinnamons (C. burmannii, C. verum, C. cassia, and C. loureiroi) using a flow injection mass spectrometric (FIMS) fingerprinting method. J Agric Food Chem. 2014 Mar 26;62(12):2516-21. doi: 10.1021/jf405580c. Epub 2014 Mar 17. PMID 24628250
- [Background] Senanayake UM, Lee TH, Wills RB. Volatile constituents of cinnamon (Cinnamomum zeylanicum) oils. Journal of agricultural and food chemistry. 1978;26(4):822-4.
- [Background] Tung YT, Chua MT, Wang SY, Chang ST. Anti-inflammation activities of essential oil and its constituents from indigenous cinnamon (Cinnamomum osmophloeum) twigs. Bioresour Technol. 2008 Jun;99(9):3908-13. doi: 10.1016/j.biortech.2007.07.050. Epub 2007 Sep 10. PMID 17826984
- [Background] Tung YT, Yen PL, Lin CY, Chang ST. Anti-inflammatory activities of essential oils and their constituents from different provenances of indigenous cinnamon (Cinnamomum osmophloeum) leaves. Pharm Biol. 2010 Oct;48(10):1130-6. doi: 10.3109/13880200903527728. PMID 20815702
- [Background] Rao PV, Gan SH. Cinnamon: a multifaceted medicinal plant. Evid Based Complement Alternat Med. 2014;2014:642942. doi: 10.1155/2014/642942. Epub 2014 Apr 10. PMID 24817901
- [Background] Litwin MS, McNaughton-Collins M, Fowler FJ Jr, Nickel JC, Calhoun EA, Pontari MA, Alexander RB, Farrar JT, O'Leary MP. The National Institutes of Health chronic prostatitis symptom index: development and validation of a new outcome measure. Chronic Prostatitis Collaborative Research Network. J Urol. 1999 Aug;162(2):369-75. doi: 10.1016/s0022-5347(05)68562-x. PMID 10411041
- [Background] Propert KJ, Litwin MS, Wang Y, Alexander RB, Calhoun E, Nickel JC, O'Leary MP, Pontari M, McNaughton-Collins M; Chronic Prostatitis Collaborative Research Network (CPCRN). Responsiveness of the National Institutes of Health Chronic Prostatitis Symptom Index (NIH-CPSI). Qual Life Res. 2006 Mar;15(2):299-305. doi: 10.1007/s11136-005-1317-1. PMID 16468084